CLINICAL TRIAL: NCT01685658
Title: Comparing the Efficacy of Intravenous Paracetamol and Ketoprofen When Treating Renal Colic in Emergency Situations: a Randomized, Bi-centric, Double-blind Controlled Trial
Brief Title: Intravenous Paracetamol Versus Ketoprofen When Treating Renal Colic in Emergency Situations
Acronym: PIVKIV
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: same study already published
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LOCAL/2012/PGC-01; 2015-002381-23 (EudraCT Number)
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Renal Colic; Acute Renal Colic
MeSH Terms: conditions — Renal Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketaprofen (Active Comparator): Patients randomized to this arm will receive intravenous ketaprofen when treating renal colic.
  Intervention: intravenous ketaprofen
  Interventions: Drug: Intravenous ketoprofen
- Paracetamol (Experimental): Patients randomized to this arm will receive intravenous paracetamol when treating renal colic.
  Intervention: intravenous paracetamol
  Interventions: Drug: Intravenous paracetamol

INTERVENTIONS:
Drug: Intravenous ketoprofen — Patients will recieve 100 mg of ketoprofen via slow intravenous perfusion. (100mg of ketoprofen powder for injection dissolved in 100 ml injectable isotonic solution)
  Arms: Ketaprofen
Drug: Intravenous paracetamol — Patients will receive 1g of paracetamol via slow intravenous perfusion. (100 ml of solution at 10mg/ml)
  Arms: Paracetamol

SUMMARY:
The main objective of this study was to demonstrate the non-inferiority of intravenous paracetamol relative to intravenous ketoprofen when treating renal colic in an emergency ward. Efficacy is measured by the change in verbal numeric scale (vns) for pain at 30 minutes.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

* To compare the efficacy (non-inferiority) of intravenous paracetamol and ketoprofen at 90 minutes (vns for pain).
* To compare both arms in terms of other administered drugs (for pain).
* To observe and compare side effects between the two arms: cutaneous manifestation, edema, bronchospasm, nausea, vomiting, headache, palpitation, chest pain, dizziness, disturbance of consciousness, dyspnea, acute retention of urine.
* To determine predictors for the use of intravenous morphine when treating renal colic.
* To compare hospitalization rates between the two groups.
* To compare patient satisfaction concerning care between the two groups (vns for satisfaction)
* To observe and compare changes towards complicated renal colic (obstructive pyelonephritis, hyperalgesia, urinary tract rupture, need for surgical drainage, sepsis, death)

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for a telephone interview at week 1
* Patient consulting at the Nîmes University Hospital emergency ward with suspicion of renal colic

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient has a contraindication for a treatment used in this study
* The patient has an allergy to ketoprofen or paracetamol, a history of gastric or intestinal ulcers, bleeding disorders, history of asthma triggered by taking ketoprofen or substances with similar activity such as other NSAIDs or aspirin
* The patient has a fever or is hemodynamically unstable, oligoanuria
* The patient presents with an initial verbal numeric pain score of 10/10.
* The patient has a history of aneurysm or aortic dissection, history of renal transplantation, history of renal or hepatic insufficiency
* The patient took paracetamol or ketoprofen 4 hours before emergency treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change in vns for pain | baseline to 30 minutes
  Verbal numeric scale ranging from 0 to 10.0.

SECONDARY OUTCOMES:
Change in vns for pain | baseline to 90 minutes
  Verbal numeric scale ranging from 0 to 10.0.
Quantity of (posology) tramadol administered | baseline (minute 0)
Quantity of (posology) tramadol administered | 30 minutes
Quantity of (posology) tramadol administered | 90 minutes
Quantity of (posology) tramadol administered | discharge from emergency ward (estimated max of 24 hours)
Quantity of (posology) phloroglucinol administered | baseline (minute 0)
Quantity of (posology) phloroglucinol administered | 30 minutes
Quantity of (posology) phloroglucinol administered | 90 minutes
Quantity of (posology) phloroglucinol administered | discharge from emergency ward (estimated max of 24 hours)
Was morphine administered? yes/no | baseline (minute 0)
Quantity of (posology) morphine administered | 30 minutes
Quantity of (posology) morphine administered | 90 minutes
Quantity of (posology) morphine administered | discharge from emergency ward (estimated max of 24 hours)
Quantity of (posology) Nefopam administered | baseline (minute 0)
Quantity of (posology) Nefopam administered | 30 minutes
Quantity of (posology) Nefopam administered | 90 minutes
Quantity of (posology) Nefopam administered | discharge from emergency ward (estimated max of 24 hours)
Quantity of (posology) Alfuzosine administered | baseline (minute 0)
Quantity of (posology) Alfuzosine administered | 30 minutes
Quantity of (posology) Alfuzosine administered | 90 minutes
Quantity of (posology) Alfuzosine administered | discharge from emergency ward (estimated max of 24 hours)
Presence/absence of complications | baseline (minute 0)
  cutaneous manifestation, edema, bronchospasm, nausea, vomiting, headache, palpitation, chest pain, dizziness, disturbance of consciousness, dyspnea, acute retention of urine
Presence/absence of complications | 30 minutes
  cutaneous manifestation, edema, bronchospasm, nausea, vomiting, headache, palpitation, chest pain, dizziness, disturbance of consciousness, dyspnea, acute retention of urine
Presence/absence of complications | 90 minutes
  cutaneous manifestation, edema, bronchospasm, nausea, vomiting, headache, palpitation, chest pain, dizziness, disturbance of consciousness, dyspnea, acute retention of urine
Presence/absence of complications | week 1
  cutaneous manifestation, edema, bronchospasm, nausea, vomiting, headache, palpitation, chest pain, dizziness, disturbance of consciousness, dyspnea, acute retention of urine
Was the patient hospitalized? yes/no | discharge from emergency ward (estimated max of 24 hours)
Was the patient hospitalized? yes/no | week 1
VNS for patient satisfaction concerning care | week 1
Evolution towards a complicated renal colic | discharge from emergency ward (estimated max of 24 hours)
  Qualitative variable with the following classes: obstructive pyelonephritis, hyperalgesia, urinary tract rupture, need for surgical drainage, sepsis, death
Evolution towards a complicated renal colic | week 1
  Qualitative variable with the following classes: obstructive pyelonephritis, hyperalgesia, urinary tract rupture, need for surgical drainage, sepsis, death

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Géraud Claret, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CH d'Alès, Alès
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes